CLINICAL TRIAL: NCT00761683
Title: Non-Interventional Study to Evaluate Effect of Zoladex In EndometrioSIS
Acronym: ESIS
Status: Terminated | Type: Observational
Why Stopped: Anticipated number of patients not achieved. All Patients recruited in the study completed all study visits.
Sponsor: AstraZeneca (Industry)
Responsible Party: Cristina Pentiuc Medical Manager, AstraZeneca
Other Study IDs: NIS-ORO-ZOL-2007/1
Record Dates: First submitted 2008-09-26; First posted 2008-09-29 (Estimated); Last update posted 2009-09-10 (Estimated); Status verified 2009-09

CONDITIONS: Endometriosis
Keywords: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients diagnosed with endometriosis

SUMMARY:
To observe the effect of goserelin 3,6mg sc depot injection by assessment of the mean percent reduction scores for symptoms: dysmenorrhoea, dyspareunia and pelvic pain; to observe the effect of goserelin 3,6mg sc depot injection by assessment of the mean percent reduction scores for pelvic tenderness and indurations; to observe the reduction in the proportion of patients requiring analgesics for the relief of pelvic pain for 6 months in patients treated with Zoladex 3.6 mg.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with endometriosis that the doctors have already decided to treat with Zoladex within the last month, before inclusion in this program, according to Romanian approved goserelin 3,6 mg

Exclusion Criteria:

* patients who have a known hypersensitivity to goserelin (Zoladex) or any of its excipients or any other GnRH analogue, pregnancy, according to Romanian approved goserelin 3,6 mg SmPC

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The programme will include the patients diagnosed with endometriosis that the doctors have already decided to treat with Zoladex within the last month, before inclusion in this program.
Sampling Method: Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2008-10

PRIMARY OUTCOMES:
Biberoglu and Bergham Scale | monthly/ at every clinic visit- 6 times for symptoms: dysmenorrhoea, dyspareunia and pelvic pain

SECONDARY OUTCOMES:
Biberoglu and Bergham Scale | twice/first and last clinic visit for pelvic tenderness and indurations

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Pentiuc, Study Director — AstraZeneca Romania
Locations (3):
- Romania (3):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Timișoara